CLINICAL TRIAL: NCT06558032
Title: Bioequivalence Study of Tamsulosin 0.4 mg Sustained Release Film Coated Tablet Produced by PT Dexa Medica in Comparison With The Comparator Drug (Harnal® Ocas 0.4 mg Prolonged Release Tablet Produced by Astellas Pharma Europe B.V., The Netherlands, Imported by PT Combiphar, Indonesia) When Administered Under Fasting Condition in Healthy Subjects
Brief Title: Bioequivalence Study of Tamsulosin 0.4 mg Sustained Release Film-coated Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BE. 827/EQL/2023
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: This was a bioequivalence study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Tamsulosin 0.4 SR PT Dexa Medica (Experimental): Tamsulosin 0.4 mg Sustained Release Tablet (produced by PT Dexa Medica, Indonesia)
  Interventions: Drug: Tamsulosin 0.4 mg Sustained Release Tablet (produced by PT Dexa Medica, Indonesia)
- Reference Harnal OCAS 0.4 mg PR Astellas, Combiphar (Active Comparator): Harnal® OCAS 0.4 mg Prolonged Release Tablet (produced by Astellas Pharma Europe B.V., The Netherlands, imported by PT Combiphar, Indonesia)
  Interventions: Drug: Harnal® OCAS 0.4 mg Prolonged Release Tablet (produced by Astellas Pharma Europe B.V., The Netherlands, imported by PT Combiphar, Indonesia)

INTERVENTIONS:
Drug: Tamsulosin 0.4 mg Sustained Release Tablet (produced by PT Dexa Medica, Indonesia) — One tablet of the test drug was given orally under fasting condition
  Arms: Test Tamsulosin 0.4 SR PT Dexa Medica
Drug: Harnal® OCAS 0.4 mg Prolonged Release Tablet (produced by Astellas Pharma Europe B.V., The Netherlands, imported by PT Combiphar, Indonesia) — One tablet of the test drug was given orally under fasting condition
  Arms: Reference Harnal OCAS 0.4 mg PR Astellas, Combiphar

SUMMARY:
This study was an open-label, randomized, single-dose, four-period, two-sequence, fully replicate study under fasting conditions which included 28 healthy adult male subjects. The objective of this study was to find out whether the bioavailability of tamsulosin 0.4 mg sustained release film coated tablet produced by PT Dexa Medica is equivalent to that of the comparator drug (Harnal® OCAS 0.4 mg Prolonged Release Tablet produced by Astellas Pharma Europe B.V., The Netherlands, imported by PT Combiphar, Indonesia) when administered under fasting condition in healthy subjects.

DETAILED DESCRIPTION:
The objective of this study was to find out whether the bioavailability of tamsulosin 0.4 mg sustained release film coated tablet produced by PT Dexa Medica is equivalent to that of the comparator drug (Harnal® OCAS 0.4 mg Prolonged Release Tablet produced by Astellas Pharma Europe B.V., The Netherlands, imported by PT Combiphar, Indonesia) when administered under fasting condition in healthy subjects. This was an open-label, randomized, single-dose, four-period, two-sequence, fully replicate study under fasting conditions which included 28 healthy adult male subjects. The participating subjects were required to have an 8 hours overnight fast and in the next morning (first day of period) were given orally the test drug (tamsulosin 0.4 mg sustained release film coated tablet produced by PT Dexa Medica) or the comparator drug (Harnal® OCAS 0.4 mg Prolonged Release Tablet produced by Astellas Pharma Europe B.V., The Netherlands, imported by PT Combiphar, Indonesia) with total 200 mL of water. The subjects' oral cavity was checked thoroughly to confirm complete medication and fluid consumption after dosing. Blood samples were drawn before taking the drug (control), and at 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 9.00, 10.00, 11.00, 12.00, 18.00, 24.00, 36.00, 48.00 and 72.00 hours after drug administration. These blood samples were used to investigate the pharmacokinetic parameters of Tamsulosin following single dose administration. The plasma concentrations of Tamsulosin were determined by using validated ultra-performance liquid chromatography with tandem mass spectroscopy detection (UPLC-MS/MS method).

ELIGIBILITY:
Inclusion Criteria:

1. Able to participate, communicate well with the investigators and willing to provide written informed consent to participate in the study.
2. Healthy male subjects with absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening and could be considered healthy based on the evaluation.
3. Aged 18 - 55 years inclusive.
4. Preferably non-smokers or smoke less than 10 cigarettes per day.
5. Body mass index within 18 to 25 kg/m2.
6. Vital signs (after 10 minutes rest) must be within the following ranges:

   * Systolic blood pressure: 110 - 129 mmHg
   * Diastolic blood pressure: 70 - 84 mmHg
   * Pulse rate: 60 - 90 bpm.
7. Willing to practice abstention or non-hormonal contraception during the study.

Exclusion Criteria:

1. History of allergy or hypersensitivity or contraindication to tamsulosin or allied drug.
2. Any major illness in the past 90 days or clinically significant ongoing chronic medical illness.
3. Presence of any clinically significant abnormal values during screening e.g. significant abnormality of liver function test (AST, ALT, alkaline phosphatase, total bilirubin, direct bilirubin ≥ 1.5 ULN), renal function test (serum creatinine concentration > 1.4 mg/dL and ureum ≥ 1.5 ULN), etc.
4. Positive Hepatitis B surface antigen (HBsAg), anti-HCV, or anti-HIV.
5. Clinically significant hematology abnormalities.
6. Clinically significant electrocardiogram (ECG) abnormalities.
7. Any surgical or medical condition (present or history) which might significantly alter the absorption, distribution, metabolism or excretion of the study drug, e.g. gastrointestinal disease including gastric or duodenal ulcers or history of gastric surgery.
8. Past history of anaphylaxis or angioedema.
9. History of drug or alcohol abuse within 12 months prior to screening for this study.
10. Participation in any clinical trial within the past 90 days calculated from the last visit until this study's first dosing day.
11. History of any bleeding or coagulative disorders.
12. Presence of difficulty in accessibility of veins in left or right arm.
13. A donation or significant blood loss within 90 days before this study's first dosing day.
14. Intake of any prescription (especially tamsulosin), non-prescription drug (including hormonal contraception), food supplements or herbal medicines within 21 days of this study's first dosing day.
15. History of orthostatic hypotension.
16. Scheduled for cataract or glaucoma surgery within 14 days after dosing.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) | 72 hours
  Area under the plasma concentration-time curve to the last observer quantifiable concentration at time t
Cmax | 72 hours
  Maximum plasma concentration

SECONDARY OUTCOMES:
AUC(0-inf) | 72 hours
  Area under the plasma concentration-time curve extrapolated to infinitive time
T1/2 | 72 hours
  Plasma half-life
Tmax | 72 hours
  Time taken to reach maximum observed plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- PT Equilab International, Jakarta, Indonesia